CLINICAL TRIAL: NCT05856838
Title: Radiofrequency Ablation in Women With Heavy Menstrual Bleeding, Procedure in an Outpatient Setting
Brief Title: NovaSure Study: Endometrial Ablation in Women With Heavy Menstrual Bleeding
Acronym: RAMBOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2023-0131
Record Dates: First submitted 2023-05-03; First posted 2023-05-12 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-01

CONDITIONS: Menstrual Bleeding, Heavy
Keywords: Menorrhagia/surgery; Endometrial Ablation Techniques; Endometrium/surgery
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NovaSure ablation (Experimental)
  Interventions: Device: NovaSure ablation

INTERVENTIONS:
Device: NovaSure ablation — Ablation of the endometrial tissue using the NovaSure device

SUMMARY:
Heavy menstrual bleeding (HMB) affects 30% of women worldwide. It negatively influences physical activity, work productivity, sexual life and overall quality of life.

In 2018, the FIGO (International Federation of Gynaecology and Obstetrics) revised its definition of AUB (FIGO-AUB system 1) and the classification of the underlying causes (FIGO-AUB system 2). It includes HMB, which is a subjective parameter and therefore patient determined. The FIGO-AUB system 2 describes the underlying causes of AUB through the acronym PALM-COEIN: Polyps, Adenomyosis, Leiomyomatosis, Malignancy, Coagulopathy, Endometrial, Iatrogenic and not otherwise specified.

The National Institute for Health and Care Excellence (NICE) guideline on HMB recommends the levonorgestrel-releasing intrauterine system (LNG-IUS) 52 mg as the treatment of first choice in women with no identified pathology, fibroids less than 3cm in diameter, which are not causing distortion of the uterine cavity, or adenomyosis. If a woman declines a LNG-IUS, non-hormonal (fibrinolytics or non-steroidal anti-inflammatory drugs (NSAIDs)) and other hormonal pharmacological treatments can be considered. If treatment is unsuccessful, the woman declines pharmacological treatment, or symptoms are severe, an endometrial ablation (EA) or hysterectomy can be an alternative option. The latter is a definitive solution, but it is an invasive option, with a risk of serious complications.

An EA is a procedure that destroys the endometrium. It aims to reduce the menstrual flow, sometimes causing amenorrhea. Initially, it was performed through hysteroscopy. Later on, second-generation devices became available. NovaSure is an example of a second-generation EA device, using a bipolar radiofrequency impedance-controlled system that evaporates endometrial tissue. The EA procedure is a minimally invasive alternative to hysterectomy. It is known to result in amenorrhea in 50% of women, with satisfaction rates between 80-96% and reported reintervention rates around 10%. Moreover, it is feasible to perform the procedure using only local anaesthesia.

The investigators aim to assess the patient acceptability and feasibility of NovaSure EA in an outpatient setting with a short observation (≤4 hours)

This observational prospective cohort study will be performed in the Ghent University Hospital (Ghent), Leuven Catholic University Hospital (Leuven) and Turnhout General Hospital (Turnhout).

The surgeon performing the procedure will be the same per institution. The duration of the study is estimated at 4 months.

DETAILED DESCRIPTION:
Eligible women will be identified by a clinician of the gynaecological department. A diagnostic hysteroscopy to rule out intrauterine abnormalities, followed by a pipelle will be done according to the local protocol of each participating centre. Written informed consent will be obtained. Participants will be asked to quantify their menstrual blood loss using the Pictorial Blood loss Assessment Chart (PBAC score) (appendix 1) before the procedure and complete the SF-36 questionnaire (appendix 2). The Novasure procedure will be scheduled at the outpatient clinic. Women will be advised to use paracetamol 1000mg and Naproxen 500mg 1 hour before the procedure. If oral NSAIDs are contra-indicated, premedication will be limited to paracetamol. During the procedure a dedicated nurse will offer personal support. Baseline characteristics (age, BMI, parity, dysmenorrhea, day of menstrual cycle at time of ablation, duration of the menstruation, use of analgesics prior to treatment and position of the uterus) will be collected. Vital parameters will be monitored during the procedure. After disinfection and speculum placement, paracervical anaesthesia (1ml of ropivacaine (Naropin) 2mg/ml) will be injected in the anterior lip of the cervix, subsequently a tenaculum will be placed. This will be followed by further paracervical infiltrations (10ml injections of ropivacaine at 3 and 9 o'clock paracervical and in both uterosacral ligaments (at 5 and 7 o'clock retrocervical)). Thereafter, a fundal infiltration will be performed through a diagnostic hysteroscopy using the Williams Cystoscopic Injection needle (Cook® Medical). Ropivacaine will be injected at 4 points in the myometrium of the fundus: 1 ml on either side of the midline and 1 ml medial to both tubal ostia. After the infiltration, speculum and tenaculum will be removed, and a 10-minute break will be taken before continuing the procedure.

After speculum placement, hysterometry will be performed and the cervix will be dilated to Hegar 8mm followed by the insertion of the NovaSure device (Classic, 8mm). A cavity assessment will be done and, if passed, ablation will start (60-90 sec). The settings of the device will be collected. After the procedure is done women can recover until they feel fit to leave (foreseen 2 to 4 hours postoperative, the time of discharge will be noted). The participants will be advised to use paracetamol 1000mg every 6 hours and Naproxen 500mg every 12 hours during 1-2 days. If oral NSAIDs were contra-indicated Tramadol will be advised. VAS scales will be used to report the intensity of the pain during the procedure and two hours after the procedure. Follow-up examination will be done 6 weeks and 3 months after the procedure. Adverse events will be recorded during the procedure and at the 6 weeks and 3 months follow-up. At the 3 months follow-up visit the following variables will be collected: patient satisfaction, symptom relief, amenorrhea rate, quality of life (SF-36), PBAC score, adverse events, additional treatment and whether they would recommend the procedure to a friend.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 35 years - ≤ 50 years
* Heavy menstrual bleeding (PBAC ≥ 150)
* Unsuccessful drug treatment, contraindication to drug treatment or rejection of drug treatment by the patient
* The absence of intra-uterine abnormalities on diagnostic hysteroscopy
* Endometrial biopsy (pipelle) is normal
* Finished childbearing

Exclusion Criteria:

* Pregnancy
* Endometritis
* Adenomyosis
* Contra-indication for local anaesthetics
* Presence of severe systemic disease (≥ASA 3)
* Previously performed endometrial ablation
* Poor understanding of Dutch language
* History of pelvic malignancy
* Presence of an intra uterine device (IUD)
* Cavity pathology (myoma, septum)
* Cavity length < 4 cm
* Each uterine incision other than conventional caesarean incision

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction assessed bij a 5-point Likert Scale | 3 months after the procedure
  Patient satisfaction of the procedure on a 5-point Likert Scale

SECONDARY OUTCOMES:
Pain assessed by VAS | During the procedure and 2 hours after the procedure
  Pain scores during and after the procedure by visual analogue score (VAS) VAS: 0-10 (0 = no pain, 1-3 = mild pain, 4-6 moderate pain, 7-9 very severe pain, 10 worst pain possible) A higher score means a worse outcome
Symptom relief assessed bij a 5-point Likert Scale | 3 months after the procedure.
  Symptom relief on a 5-point Likert Scale
  1. Very unsatisfied
  2. A little bit unsatisfied
  3. Neutral
  4. Satisfied
  5. Very satisfied
  A high score means a good outcome.
Amenorrhea rate | at 6 weeks and 3 months after the procedure.
  Frequency of the menstruation cycle
Menstrual blood loss | 1 month before and 3 months after the procedure.
  quantified by the Pictorial Blood loss Assessment Chart (PBAC score) A high score means more bloodloss (maximum 150 score).
Health related quality of life assessment | 1 month before and 3 months after the procedure.
  Health related quality of life measured by the SF-36 questionnaire
Adverse events | During and up to 6 weeks and 3 months after the procedure.
  Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the investigational medical device.
  A serious adverse event is any untoward medical occurrence or effect that
  1. results in death;
  2. is life threatening (at the time of the event);
  3. requires hospitalization or prolongation of existing inpatients' hospitalization;
  4. results in persistent or significant disability or incapacity;
  5. any other important medical event that did not result in any of the outcomes listed above due to medical or surgical intervention but could have been based upon appropriate judgement by the investigator. An elective hospital admission will not be considered as a serious adverse event.
Any additional treatment needed after NovaSure procedure | 3 months after the procedure.
  Non-hormonal medication, hormonal medication (oral combination pil, IUD), surgery (hysterectomy for example).
Recommendation to a friend | 3 months after the procedure.
  Whether they would recommend the procedure to a friend (Yes/No) at 3 months after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No